CLINICAL TRIAL: NCT06075108
Title: P-KIDs CARE: An Intervention to Address Health Systems Delays to Care for Injured Children in Tanzania
Brief Title: The P-KIDs CARE Health Systems Intervention in Tanzania
Acronym: P-KIDs CARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Kilimanjaro Christian Medical Centre, Tanzania (Other); Kilimanjaro Clinical Research Institute (Other)
Responsible Party: Principal Investigator, Elizabeth M. Keating, MD, MSPH - Assistant Professor, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB_00169039
Record Dates: First submitted 2023-09-12; First posted 2023-10-10 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Accidental Injuries; Global Child Health; Pediatric Emergency Medicine; Public Health System Research; Health Care Providers; Implementation Science
Keywords: Accidental Injuries; Global Child Health; Pediatric Emergency Medicine; Health Care Providers; Public Health System Research; Implementation Science
MeSH Terms: conditions — Accidental Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- P-KIDs CARE (Other): The P-KIDs CARE intervention will include two components: 1) the World Health Organization (WHO) Basic Emergency Care Course for training on patient assessment and stabilization, and 2) a decision support tool which integrates adaptation of two evidence-based tools: a) the Pediatric Resuscitation and Trauma Outcome model for mortality risk assessment, and 3) the Field Triage Decision Scheme to assist with timely referral decisions. WHO Basic Emergency Care Course includes modules delivered via PowerPoint with hands-on training components. The decision support tool will be online with checkboxes that healthcare providers can cross as they fill it out in real time. The team will adapt the tool for use in Northern Tanzania, with particular attention to local contextual and cultural factors.
  Interventions: Other: P-KIDs CARE

INTERVENTIONS:
Other: P-KIDs CARE — The P-KIDs CARE intervention will include two components: 1) the World Health Organization (WHO) Basic Emergency Care Course for training on patient assessment and stabilization, and 2) a decision support tool which integrates adaptation of two evidence-based tools: a) the Pediatric Resuscitation and Trauma Outcome model for mortality risk assessment, and 3) the Field Triage Decision Scheme to assist with timely referral decisions. WHO Basic Emergency Care Course includes modules delivered via PowerPoint with hands-on training components. The decision support tool will be online with checkboxes that healthcare providers can cross as they fill it out in real time. The team will adapt the tool for use in Northern Tanzania, with particular attention to local contextual and cultural factors.
  Other Names: Health systems intervention

SUMMARY:
The objective of the proposed research is to develop and pilot a locally-relevant, multicomponent intervention to streamline the triage process (e.g. patient assessment, stabilization, and disposition) for pediatric injury patients in Tanzania. This health systems intervention will work at the first level of medical contact (e.g., health center and district hospital), in order to facilitate timely disposition and referrals, and subsequently decrease time to definitive care. The proposed study has three aims: 1) With a mixed methods approach, describe the barriers to pediatric injury care at the first medical contact; 2) Iteratively develop the P-KIDs CARE intervention using a nominal group technique and conduct a pre-implementation assessment and refinement; 3) Pilot the P-KIDs CARE intervention and perform an implementation-focused formative evaluation. The proposed study focuses on pediatric injury patients and the family members and healthcare providers that care for them in Kilimanjaro, Tanzania. The investigators will recruit pediatric injury patients, family members, and healthcare providers from 2 health facilities in the Kilimanjaro Region.

DETAILED DESCRIPTION:
In Aim 1, the investigators will conduct formative research to inform development of the P-KIDs CARE intervention. The investigators will enroll 100 children into the pediatric injury registry and conduct capacity assessments of the two study facilities using the WHO Health Emergency Unit Assessment Tool. The investigators will conduct in-depth interviews (IDIs) with 15 family members of pediatric injury patients who were referred and made it to Kilimanjaro Christian Medical Centre (KCMC), and 15 family members of pediatric injury patients who were referred but did not make it to KCMC. The investigators will conduct 2 focus group discussions (FGDs) with approximately 10-15 healthcare providers of pediatric injury patients at each of the 2 the study facilities. In Aim 2, the investigators will use this formative data to develop the P-KIDs CARE intervention during a 2-day intervention development workshop with an interdisciplinary study team. The investigators will then perform a pre-implementation assessment and refinement by convening focus group discussions with healthcare providers and a community-engaged panel. This step will enable us to obtain feedback and refine the intervention. In Aim 3, the investigators will pilot the intervention in 2 study facilities in the Kilimanjaro Region. The investigators anticipate 10 total healthcare providers will be enrolled across the 2 study facilities. The investigators expect to enroll approximately 200 pediatric injury patients, 100 in the pre-intervention period and 100 in the post-intervention period. The investigators will conduct post-surveys and exit interviews for healthcare providers using the intervention, assessing implementation outcomes including feasibility, healthcare provider acceptability, and fidelity. The investigators will also conduct interviews with family members of 12 patients referred to KCMC and 12 patients not referred, assessing acceptability and satisfaction with the disposition decision. The investigators will also collect patient-level, potential trial outcomes including time from first care to definitive care, disposition, morbidity, and mortality. The primary outcome will be mortality. The second outcomes will be time to definitive care, disposition, and morbidity. While not powered to determine effect size, the investigators hope that preliminary analysis will suggest a signal of difference between groups.

ELIGIBILITY:
Inclusion Criteria:

* AIM 1 (mixed methods research)

  1. Enroll into the pediatric injury registry all pediatric (<18 years old) patients seeking care at one of the study health facilities for an acute injury.
  2. The investigators will conduct in-depth interviews with the following group: Family members of a pediatric injury patients seeking care at the study facilities.
  3. The investigators will conduct focus group discussions with the following group: Health care providers providing care to pediatric injury patients at the study facilities.
* AIM 2 (develop intervention)

  1. The investigators will hold a 2-day intervention development workshop with the interdisciplinary study team.
  2. The investigators will conduct focus group discussions with the following groups:

     1. Health care providers providing care to pediatric injury patients at the study health facilities
     2. A community-engaged panel including family members of pediatric injury patients
* AIM 3 (pilot intervention)

  1. The investigators will enroll into the pediatric injury registry all pediatric (<18 years old) patients seeking care at one of the study health facilities for an acute injury.
  2. The investigators will conduct surveys and exit interviews with the following groups:

     1. Health care providers providing care to pediatric injury patients at the study health facilities.
     2. Family members of pediatric injury patients.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 284 (Estimated)
Dates: Start 2024-08-05 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | Baseline (baseline data collection over 1 year in study years 1-2) and post intervention implementation (data collection over 1 year in study year 4); two data collection periods will be separated by 1.5 years
  Mortality as binary outcome variable

SECONDARY OUTCOMES:
Time from patients' injury to definitive care at Kilimanjaro Christian Medical Center (KCMC) measured via a pediatric injury registry | Baseline (baseline data collection over 1 year in study years 1-2) and post intervention implementation (data collection over 1 year in study year 4); two data collection periods will be separated by 1.5 years
  Time from patient's injury to definitive care at KCMC as continuous variable measured via a pediatric injury registry
Patient disposition | Baseline (baseline data collection over 1 year in study years 1-2) and post intervention implementation (data collection over 1 year in study year 4); two data collection periods will be separated by 1.5 years
  Location of patient disposition after care at health facility with options including: discharge home, admission to health facility, transfer to other health facility
Patient morbidity as measured by the Glasgow Outcomes Scale-Extended Pediatrics | Baseline (baseline data collection over 1 year in study years 1-2) and post intervention implementation (data collection over 1 year in study year 4); two data collection periods will be separated by 1.5 years
  Patient morbidity as measured by the Glasgow Outcomes Scale-Extended Pediatrics; binary variable with 1-2 indicating good outcome, 3-8 indicating poor outcome

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth M. Keating, MD, Principal Investigator — University of Utah
Locations (1):
- Kilimanjaro Christian Medical Centre, Moshi, Tanzania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Keating EM, Nget P, Kea S, Kuong S, Daly L, Phearom S, Enders F, Cheryk LA, Topazian M, Fischer PR, Kumar V. Thiamine deficiency in tachypnoeic Cambodian infants. Paediatr Int Child Health. 2015;35(4):312-8. doi: 10.1080/20469047.2015.1109226. Epub 2014 Oct 27. PMID 26744155
- [Background] Keating EM, Lukolyo H, Crouse HL, Pitt MB, St Clair N, Butteris S. Socially Awkward Abroad: A Call for Social Media Policies in Residencies that Offer Global Health Electives. Am J Trop Med Hyg. 2018 Nov;99(5):1275-1282. doi: 10.4269/ajtmh.18-0501. PMID 30226146
- [Background] Keating EM, Lukolyo H, Rees CA, Dziuban EJ, Ferris MG, Schutze GE, Marton SA. Beyond the learning curve: length of global health electives. Int J Med Educ. 2016 Sep 11;7:295-6. doi: 10.5116/ijme.57c1.4e07. No abstract available. PMID 27614032
- [Background] Lukolyo H, Rees CA, Keating EM, Swamy P, Schutze GE, Marton S, Turner TL. Perceptions and Expectations of Host Country Preceptors of Short-Term Learners at Four Clinical Sites in Sub-Saharan Africa. Acad Pediatr. 2016 May-Jun;16(4):387-93. doi: 10.1016/j.acap.2015.11.002. Epub 2015 Nov 12. PMID 26581780
- [Background] Rees CA, Keating EM, Lukolyo H, Danysh HE, Scheurer ME, Mehta PS, Lubega J, Slone JS; Baylor Pediatric HIV-Related Malignancy Consortium. Mapping the Epidemiology of Kaposi Sarcoma and Non-Hodgkin Lymphoma Among Children in Sub-Saharan Africa: A Review. Pediatr Blood Cancer. 2016 Aug;63(8):1325-31. doi: 10.1002/pbc.26021. Epub 2016 Apr 15. PMID 27082516
- [Background] Rees CA, Keating EM, Lukolyo H, Swamy P, Turner TL, Marton S, Sanders J, Mohapi EQ, Kazembe PN, Schutze GE. Host clinical preceptors' perceptions of professionalism among learners completing global health electives. Int J Med Educ. 2018 Jul 27;9:206-212. doi: 10.5116/ijme.5b40.6e4b. PMID 30055101
- [Background] Rees CA, Lukolyo H, Keating EM, Dearden KA, Luboga SA, Schutze GE, Kazembe PN. Authorship in paediatric research conducted in low- and middle-income countries: parity or parasitism? Trop Med Int Health. 2017 Nov;22(11):1362-1370. doi: 10.1111/tmi.12966. Epub 2017 Sep 20. PMID 28857354
- [Background] Slusher TM, Zamora TG, Appiah D, Stanke JU, Strand MA, Lee BW, Richardson SB, Keating EM, Siddappa AM, Olusanya BO. Burden of severe neonatal jaundice: a systematic review and meta-analysis. BMJ Paediatr Open. 2017 Nov 25;1(1):e000105. doi: 10.1136/bmjpo-2017-000105. eCollection 2017. PMID 29637134
- [Background] Keating EM, Sanders J, Ngo K, Mohapi EQ, Mandalakas AM. Development of a Tool for Health Screening and Assessment in Orphanages in Lesotho. Am J Trop Med Hyg. 2019 May;100(5):1290-1293. doi: 10.4269/ajtmh.18-0853. PMID 30915954
- [Background] Lukolyo H, Keating EM, Rees CA. Creating a collaborative peer writing group during residency. Med Educ Online. 2019 Dec;24(1):1563421. doi: 10.1080/10872981.2018.1563421. PMID 30813852
- [Background] Rees CA, Keating EM, Dearden KA, Haq H, Robison JA, Kazembe PN, Bourgeois FT, Niescierenko M. Importance of authorship and inappropriate authorship assignment in paediatric research in low- and middle-income countries. Trop Med Int Health. 2019 Oct;24(10):1229-1242. doi: 10.1111/tmi.13295. Epub 2019 Aug 21. PMID 31374140
- [Background] Rees CA, Keating EM, Dearden KA, Haq H, Robison JA, Kazembe PN, Bourgeois FT, Niescierenko M. Improving Pediatric Academic Global Health Collaborative Research and Agenda Setting: A Mixed-Methods Study. Am J Trop Med Hyg. 2020 Mar;102(3):649-657. doi: 10.4269/ajtmh.19-0555. PMID 31933470
- [Background] Keating EM, Chiume M, Fitzgerald E, Mgusha Y, Mvalo T, Fino N, Crouse HL, Eckerle M, Gorman K, Ciccone EJ, Airewele G, Robison JA. Blood transfusion and mortality in children with severe anaemia in a malaria-endemic region. Paediatr Int Child Health. 2021 May;41(2):129-136. doi: 10.1080/20469047.2021.1881270. Epub 2021 Apr 19. PMID 33874852
- [Background] Keating EM, Robison JA, Chiume M, Taddie M, VanDerslice JA, Benson LS, Fitzgerald E, Crouse HL, Eckerle MD, Ciccone EJ, Porucznik CA. Relationship between distance of referring facilities and haemoglobin change in children in Malawi. Paediatr Int Child Health. 2021 Nov;41(4):253-261. doi: 10.1080/20469047.2022.2044674. Epub 2022 Mar 1. PMID 35230927
- [Background] Keating EM, Price RR, Robison JA. Paediatric trauma epidemic: a call to action. BMJ Paediatr Open. 2019 Aug 1;3(1):e000532. doi: 10.1136/bmjpo-2019-000532. eCollection 2019. No abstract available. PMID 31423470
- [Background] Keating EM, Sakita F, Mmbaga BT, Amiri I, Nkini G, Rent S, Fino N, Young B, Staton CA, Watt MH. Three delays model applied to pediatric injury care seeking in Northern Tanzania: A mixed methods study. PLOS Glob Public Health. 2022 Aug 25;2(8):e0000657. doi: 10.1371/journal.pgph.0000657. eCollection 2022. PMID 36962759
- [Background] Peden M, Oyegbite K, Ozanne-Smith J, Hyder AA, Branche C, Rahman AKMF, Rivara F, Bartolomeos K, editors. World Report on Child Injury Prevention. Geneva: World Health Organization; 2008. Available from http://www.ncbi.nlm.nih.gov/books/NBK310641/ PMID 26269872
- [Background] GBD 2017 Causes of Death Collaborators. Global, regional, and national age-sex-specific mortality for 282 causes of death in 195 countries and territories, 1980-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2018 Nov 10;392(10159):1736-1788. doi: 10.1016/S0140-6736(18)32203-7. Epub 2018 Nov 8. PMID 30496103
- [Background] Abdur-Rahman LO, van As AB, Rode H. Pediatric trauma care in Africa: the evolution and challenges. Semin Pediatr Surg. 2012 May;21(2):111-5. doi: 10.1053/j.sempedsurg.2012.01.003. PMID 22475116
- [Background] St-Louis E, Petroze R, Baird R, Razek T, Poenaru D, Calland JF, Byiringiro JC, Ntaganda E. Calibration and validation of the pediatric resuscitation and trauma outcome model among injured children in Rwanda. J Pediatr Surg. 2020 Nov;55(11):2510-2516. doi: 10.1016/j.jpedsurg.2020.01.056. Epub 2020 Feb 19. PMID 32151404
- [Background] Botchey IM Jr, Hung YW, Bachani AM, Saidi H, Paruk F, Hyder AA. Understanding patterns of injury in Kenya: Analysis of a trauma registry data from a National Referral Hospital. Surgery. 2017 Dec;162(6S):S54-S62. doi: 10.1016/j.surg.2017.02.016. Epub 2017 Apr 21. PMID 28438334
- [Background] Boyd DR, Cowley RA. Comprehensive regional trauma/emergency medical services (EMS) delivery systems: the United States experience. World J Surg. 1983 Jan;7(1):149-57. doi: 10.1007/BF01655923. No abstract available. PMID 6837054
- [Background] Rogers FB, Rittenhouse KJ, Gross BW. The golden hour in trauma: dogma or medical folklore? Injury. 2015 Apr;46(4):525-7. doi: 10.1016/j.injury.2014.08.043. Epub 2014 Sep 16. No abstract available. PMID 25262329
- [Background] Mock C, Abantanga F, Goosen J, Joshipura M, Juillard C. Strengthening care of injured children globally. Bull World Health Organ. 2009 May;87(5):382-9. doi: 10.2471/blt.08.057059. PMID 19551257
- [Background] Wisborg T, Montshiwa TR, Mock C. Trauma research in low- and middle-income countries is urgently needed to strengthen the chain of survival. Scand J Trauma Resusc Emerg Med. 2011 Oct 24;19:62. doi: 10.1186/1757-7241-19-62. PMID 22024376
- [Background] Sa'avu M, Duke T, Matai S. Improving paediatric and neonatal care in rural district hospitals in the highlands of Papua New Guinea: a quality improvement approach. Paediatr Int Child Health. 2014 May;34(2):75-83. doi: 10.1179/2046905513Y.0000000081. Epub 2013 Dec 6. PMID 24621233
- [Background] Jin J, Akau'ola S, Yip CH, Nthumba P, Ameh EA, de Jonge S, Mehes M, Waiqanabete I, Henry J, Hill A; International Society of Surgery (ISS) and the G4 Alliance International Standards and Guidelines for Quality Safe Surgery and Anesthesia (ISG-QSSA) Group. Effectiveness of Quality Improvement Processes, Interventions, and Structure in Trauma Systems in Low- and Middle-Income Countries: A Systematic Review and Meta-analysis. World J Surg. 2021 Jul;45(7):1982-1998. doi: 10.1007/s00268-021-06065-9. Epub 2021 Apr 9. PMID 33835217
- [Background] Husum H, Gilbert M, Wisborg T, Van Heng Y, Murad M. Rural prehospital trauma systems improve trauma outcome in low-income countries: a prospective study from North Iraq and Cambodia. J Trauma. 2003 Jun;54(6):1188-96. doi: 10.1097/01.TA.0000073609.12530.19. PMID 12813342
- [Background] Whitaker J, Nepogodiev D, Leather A, Davies J. Assessing barriers to quality trauma care in low and middle-income countries: A Delphi study. Injury. 2020 Feb;51(2):278-285. doi: 10.1016/j.injury.2019.12.035. Epub 2019 Dec 21. PMID 31883865
- [Background] Kironji AG, Hodkinson P, de Ramirez SS, Anest T, Wallis L, Razzak J, Jenson A, Hansoti B. Identifying barriers for out of hospital emergency care in low and low-middle income countries: a systematic review. BMC Health Serv Res. 2018 Apr 19;18(1):291. doi: 10.1186/s12913-018-3091-0. PMID 29673360
- [Background] Chokotho L, Mulwafu W, Singini I, Njalale Y, Maliwichi-Senganimalunje L, Jacobsen KH. First Responders and Prehospital Care for Road Traffic Injuries in Malawi. Prehosp Disaster Med. 2017 Feb;32(1):14-19. doi: 10.1017/S1049023X16001175. Epub 2016 Dec 7. PMID 27923422
- [Background] Gyedu A, Baah EG, Boakye G, Ohene-Yeboah M, Otupiri E, Stewart BT. Quality of referrals for elective surgery at a tertiary care hospital in a developing country: an opportunity for improving timely access to and cost-effectiveness of surgical care. Int J Surg. 2015 Mar;15:74-8. doi: 10.1016/j.ijsu.2015.01.033. Epub 2015 Feb 4. PMID 25659222
- [Background] Mock CN, Donkor P, Gawande A, Jamison DT, Kruk ME, Debas HT; DCP3 Essential Surgery Author Group. Essential surgery: key messages from Disease Control Priorities, 3rd edition. Lancet. 2015 May 30;385(9983):2209-19. doi: 10.1016/S0140-6736(15)60091-5. Epub 2015 Feb 5. PMID 25662414
- [Background] Thomas D, Mujugira A, Ortblad K, Namanda S, Kibuuka J, Nakitende M, Nambi F, Nakabugo L, Scoville C, Muwonge T, Heffron R. A pragmatic approach to identifying implementation barriers and facilitators for a novel pre-exposure prophylaxis (PrEP) delivery model at public facilities in urban Uganda. Implement Sci Commun. 2022 Jan 28;3(1):7. doi: 10.1186/s43058-022-00254-w. PMID 35090560
- [Background] Michaud-Letourneau I, Gayard M, Njoroge B, Agabiirwe CN, Luwangula AK, McGough L, Mwangi A, Pelto G, Tumilowicz A, Pelletier DL. Operationalizing Implementation Science in Nutrition: The Implementation Science Initiative in Kenya and Uganda. Curr Dev Nutr. 2021 Nov 29;6(1):nzab146. doi: 10.1093/cdn/nzab146. eCollection 2022 Jan. PMID 35047720
- [Background] Le PD, Eschliman EL, Grivel MM, Tang J, Cho YG, Yang X, Tay C, Li T, Bass J, Yang LH. Barriers and facilitators to implementation of evidence-based task-sharing mental health interventions in low- and middle-income countries: a systematic review using implementation science frameworks. Implement Sci. 2022 Jan 12;17(1):4. doi: 10.1186/s13012-021-01179-z. PMID 35022081
- [Background] Turner MW, Bogdewic S, Agha E, Blanchard C, Sturke R, Pettifor A, Salisbury K, Marques AH, Excellent ML, Rajagopal N, Ramaswamy R. Learning needs assessment for multi-stakeholder implementation science training in LMIC settings: findings and recommendations. Implement Sci Commun. 2021 Dec 4;2(1):134. doi: 10.1186/s43058-021-00238-2. PMID 34863314
- [Background] Brown S, Leavy JE, Jancey J. Implementation of GeneXpert for TB Testing in Low- and Middle-Income Countries: A Systematic Review. Glob Health Sci Pract. 2021 Sep 30;9(3):698-710. doi: 10.9745/GHSP-D-21-00121. Print 2021 Sep 30. PMID 34593592
- [Background] Taylor Salisbury T, Kohrt BA, Bakolis I, Jordans MJ, Hull L, Luitel NP, McCrone P, Sevdalis N, Pokhrel P, Carswell K, Ojagbemi A, Green EP, Chowdhary N, Kola L, Lempp H, Dua T, Milenova M, Gureje O, Thornicroft G. Adaptation of the World Health Organization Electronic Mental Health Gap Action Programme Intervention Guide App for Mobile Devices in Nepal and Nigeria: Protocol for a Feasibility Cluster Randomized Controlled Trial. JMIR Res Protoc. 2021 Jun 15;10(6):e24115. doi: 10.2196/24115. PMID 34128819
- [Background] Ojo T, Kabasele L, Boyd B, Enechukwu S, Ryan N, Gyamfi J, Peprah E. The Role of Implementation Science in Advancing Resource Generation for Health Interventions in Low- and Middle-Income Countries. Health Serv Insights. 2021 Mar 15;14:1178632921999652. doi: 10.1177/1178632921999652. eCollection 2021. PMID 33795935
- [Background] Kumar M, Huang KY, Othieno C, Wamalwa D, Hoagwood K, Unutzer J, Saxena S, Petersen I, Njuguna S, Amugune B, Gachuno O, Ssewamala F, McKay M. Implementing combined WHO mhGAP and adapted group interpersonal psychotherapy to address depression and mental health needs of pregnant adolescents in Kenyan primary health care settings (INSPIRE): a study protocol for pilot feasibility trial of the integrated intervention in LMIC settings. Pilot Feasibility Stud. 2020 Sep 22;6:136. doi: 10.1186/s40814-020-00652-8. eCollection 2020. PMID 32974045
- [Background] Peiffer-Smadja N, Poda A, Ouedraogo AS, Guiard-Schmid JB, Delory T, Le Bel J, Bouvet E, Lariven S, Jeanmougin P, Ahmad R, Lescure FX. Paving the Way for the Implementation of a Decision Support System for Antibiotic Prescribing in Primary Care in West Africa: Preimplementation and Co-Design Workshop With Physicians. J Med Internet Res. 2020 Jul 20;22(7):e17940. doi: 10.2196/17940. PMID 32442155
- [Background] Romani ED, Siddharthan T, Lovaton N, Alvitez-Luna CC, Flores-Flores O, Pollard SL. Implementation of an intervention to improve the adoption of asthma self-management practices in Peru: Asthma Implementation Research (AIRE) randomized trial study protocol. Trials. 2020 May 4;21(1):377. doi: 10.1186/s13063-020-4207-5. PMID 32366314
- [Background] Means AR, Kemp CG, Gwayi-Chore MC, Gimbel S, Soi C, Sherr K, Wagenaar BH, Wasserheit JN, Weiner BJ. Evaluating and optimizing the consolidated framework for implementation research (CFIR) for use in low- and middle-income countries: a systematic review. Implement Sci. 2020 Mar 12;15(1):17. doi: 10.1186/s13012-020-0977-0. PMID 32164692
- [Background] Keating EM, Mitao M, Kozhumam A, Souza JV, Anthony CS, Costa DB, Staton CA, Mmbaga BT, Vissoci JRN. Validation of the Pediatric Resuscitation and Trauma Outcome (PRESTO) model in injury patients in Tanzania. BMJ Open. 2023 Apr 5;13(4):e070747. doi: 10.1136/bmjopen-2022-070747. PMID 37019480
- [Background] Sasser SM, Hunt RC, Faul M, Sugerman D, Pearson WS, Dulski T, Wald MM, Jurkovich GJ, Newgard CD, Lerner EB; Centers for Disease Control and Prevention (CDC). Guidelines for field triage of injured patients: recommendations of the National Expert Panel on Field Triage, 2011. MMWR Recomm Rep. 2012 Jan 13;61(RR-1):1-20. PMID 22237112
- [Background] Bhaumik S, Hannun M, Dymond C, DeSanto K, Barrett W, Wallis LA, Mould-Millman NK. Prehospital triage tools across the world: a scoping review of the published literature. Scand J Trauma Resusc Emerg Med. 2022 Apr 27;30(1):32. doi: 10.1186/s13049-022-01019-z. PMID 35477474
- [Background] Ardolino A, Cheung CR, Lawrence T, Bouamra O, Lecky F, Berry K, Lyttle M, Roland D, Koralage N, Issa S, Chaudhary A, Maconochie I; PERUKI group. The accuracy of existing prehospital triage tools for injured children in England: an analysis using emergency department data. Emerg Med J. 2015 May;32(5):397-400. doi: 10.1136/emermed-2013-203251. Epub 2014 Apr 8. PMID 24714672
- [Background] Lerner EB, Cushman JT, Drendel AL, Badawy M, Shah MN, Guse CE, Cooper A. Effect of the 2011 Revisions to the Field Triage Guidelines on Under- and Over-Triage Rates for Pediatric Trauma Patients. Prehosp Emerg Care. 2017 Jul-Aug;21(4):456-460. doi: 10.1080/10903127.2017.1300717. Epub 2017 May 10. PMID 28489471
- [Background] Baker A, Cornwell P, Gustafsson L, Stewart C, Lannin NA. Developing tailored theoretically informed goal-setting interventions for rehabilitation services: a co-design approach. BMC Health Serv Res. 2022 Jun 22;22(1):811. doi: 10.1186/s12913-022-08047-6. PMID 35733190
- [Background] Al-Mondhiry J, D'Ambruoso S, Pietras C, Strouse T, Benzeevi D, Arevian AC, Wells KB. Co-created Mobile Apps for Palliative Care Using Community-Partnered Participatory Research: Development and Usability Study. JMIR Form Res. 2022 Jun 23;6(6):e33849. doi: 10.2196/33849. PMID 35737441
- [Background] Brusco NK, Atkinson V, Woods J, Myles PS, Hodge A, Jones C, Lloyd D, Rovtar V, Clifford AM, Morris ME. Implementing PROMS for elective surgery patients: feasibility, response rate, degree of recovery and patient acceptability. J Patient Rep Outcomes. 2022 Jul 7;6(1):73. doi: 10.1186/s41687-022-00483-6. PMID 35798915
- [Background] Toomey CM, Kennedy N, MacFarlane A, Glynn L, Forbes J, Skou ST, Roos EM. Implementation of clinical guidelines for osteoarthritis together (IMPACT): protocol for a participatory health research approach to implementing high value care. BMC Musculoskelet Disord. 2022 Jul 5;23(1):643. doi: 10.1186/s12891-022-05599-w. PMID 35790924
- [Background] McLachlan HL, Newton M, McLardie-Hore FE, McCalman P, Jackomos M, Bundle G, Kildea S, Chamberlain C, Browne J, Ryan J, Freemantle J, Shafiei T, Jacobs SE, Oats J, Blow N, Ferguson K, Gold L, Watkins J, Dell M, Read K, Hyde R, Matthews R, Forster DA. Translating evidence into practice: Implementing culturally safe continuity of midwifery care for First Nations women in three maternity services in Victoria, Australia. EClinicalMedicine. 2022 May 4;47:101415. doi: 10.1016/j.eclinm.2022.101415. eCollection 2022 May. PMID 35747161
- [Background] Burstein B, Fauteux-Lamarre E, As AB. Increased morbidity associated with weekend paediatric road traffic injuries: 10-year analysis of trauma registry data. Injury. 2016 Jun;47(6):1236-41. doi: 10.1016/j.injury.2016.02.021. Epub 2016 Mar 3. PMID 27084114
- [Background] Traynor MD Jr, St Louis E, Hernandez MC, Alsayed AS, Klinkner DB, Baird R, Poenaru D, Kong VY, Moir CR, Zielinski MD, Laing GL, Bruce JL, Clarke DL. Comparison of the Pediatric Resuscitation and Trauma Outcome (PRESTO) Model and Pediatric Trauma Scoring Systems in a Middle-Income Country. World J Surg. 2020 Aug;44(8):2518-2525. doi: 10.1007/s00268-020-05512-3. PMID 32314007
- [Background] Bradshaw CJ, Bandi AS, Muktar Z, Hasan MA, Chowdhury TK, Banu T, Hailemariam M, Ngu F, Croaker D, Bankole R, Sholadoye T, Olaomi O, Ameh E, Di Cesare A, Leva E, Ringo Y, Abdur-Rahman L, Salama R, Elhalaby E, Perera H, Parsons C, Cleeve S, Numanoglu A, Van As S, Sharma S, Lakhoo K. International Study of the Epidemiology of Paediatric Trauma: PAPSA Research Study. World J Surg. 2018 Jun;42(6):1885-1894. doi: 10.1007/s00268-017-4396-6. PMID 29282513
- [Background] Petroze RT, Martin AN, Ntaganda E, Kyamanywa P, St-Louis E, Rasmussen SK, Calland JF, Byiringiro JC. Epidemiology of paediatric injuries in Rwanda using a prospective trauma registry. BJS Open. 2020 Feb;4(1):78-85. doi: 10.1002/bjs5.50222. Epub 2019 Nov 17. PMID 32011812
- [Background] Aluisio AR, Waheed S, Cameron P, Hess J, Jacob ST, Kissoon N, Levine AC, Mian A, Ramlakhan S, Sawe HR, Razzak J. Clinical emergency care research in low-income and middle-income countries: opportunities and challenges. BMJ Glob Health. 2019 Jul 29;4(Suppl 6):e001289. doi: 10.1136/bmjgh-2018-001289. eCollection 2019. PMID 31406600
- [Background] Millum J, Beecroft B, Hardcastle TC, Hirshon JM, Hyder AA, Newberry JA, Saenz C. Emergency care research ethics in low-income and middle-income countries. BMJ Glob Health. 2019 Jul 29;4(Suppl 6):e001260. doi: 10.1136/bmjgh-2018-001260. eCollection 2019. PMID 31406598
- [Background] Moresky RT, Razzak J, Reynolds T, Wallis LA, Wachira BW, Nyirenda M, Carlo WA, Lin J, Patel S, Bhoi S, Risko N, Wendle LA, Calvello Hynes EJ; National Institute of Health Fogarty International Center convened the Collaborative on Enhancing Emergency Care Research in LMICs (CLEER). Advancing research on emergency care systems in low-income and middle-income countries: ensuring high-quality care delivery systems. BMJ Glob Health. 2019 Jul 29;4(Suppl 6):e001265. doi: 10.1136/bmjgh-2018-001265. eCollection 2019. PMID 31406599
- [Background] Mowafi H, Ngaruiya C, O'Reilly G, Kobusingye O, Kapil V, Rubiano A, Ong M, Puyana JC, Rahman AF, Jooma R, Beecroft B, Razzak J. Emergency care surveillance and emergency care registries in low-income and middle-income countries: conceptual challenges and future directions for research. BMJ Glob Health. 2019 Jul 29;4(Suppl 6):e001442. doi: 10.1136/bmjgh-2019-001442. eCollection 2019. PMID 31406601
- [Background] Razzak J, Beecroft B, Brown J, Hargarten S, Anand N. Emergency care research as a global health priority: key scientific opportunities and challenges. BMJ Glob Health. 2019 Jul 29;4(Suppl 6):e001486. doi: 10.1136/bmjgh-2019-001486. eCollection 2019. PMID 31406602
- [Background] Kruk ME, Gage AD, Arsenault C, Jordan K, Leslie HH, Roder-DeWan S, Adeyi O, Barker P, Daelmans B, Doubova SV, English M, Garcia-Elorrio E, Guanais F, Gureje O, Hirschhorn LR, Jiang L, Kelley E, Lemango ET, Liljestrand J, Malata A, Marchant T, Matsoso MP, Meara JG, Mohanan M, Ndiaye Y, Norheim OF, Reddy KS, Rowe AK, Salomon JA, Thapa G, Twum-Danso NAY, Pate M. High-quality health systems in the Sustainable Development Goals era: time for a revolution. Lancet Glob Health. 2018 Nov;6(11):e1196-e1252. doi: 10.1016/S2214-109X(18)30386-3. Epub 2018 Sep 5. No abstract available. PMID 30196093
- [Background] Whitaker J, O'Donohoe N, Denning M, Poenaru D, Guadagno E, Leather AJM, Davies JI. Assessing trauma care systems in low-income and middle-income countries: a systematic review and evidence synthesis mapping the Three Delays framework to injury health system assessments. BMJ Glob Health. 2021 May;6(5):e004324. doi: 10.1136/bmjgh-2020-004324. PMID 33975885
- [Background] Keith RE, Crosson JC, O'Malley AS, Cromp D, Taylor EF. Using the Consolidated Framework for Implementation Research (CFIR) to produce actionable findings: a rapid-cycle evaluation approach to improving implementation. Implement Sci. 2017 Feb 10;12(1):15. doi: 10.1186/s13012-017-0550-7. PMID 28187747
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Beers SR, Wisniewski SR, Garcia-Filion P, Tian Y, Hahner T, Berger RP, Bell MJ, Adelson PD. Validity of a pediatric version of the Glasgow Outcome Scale-Extended. J Neurotrauma. 2012 Apr 10;29(6):1126-39. doi: 10.1089/neu.2011.2272. Epub 2012 Apr 10. PMID 22220819
- [Background] Mann M, Musabyemariya I, Harding L, Braxley B. Using Patient-Reported Outcome Measures to Promote Patient-Centered Practice: Building Capacity Among Pediatric Physiotherapists in Rwanda. Glob Health Sci Pract. 2020 Sep 30;8(3):596-605. doi: 10.9745/GHSP-D-19-00408. Print 2020 Sep 30. PMID 33008866
- [Background] Chavula C, Pigoga JL, Kafwamfwa M, Wallis LA. Cross-sectional evaluation of emergency care capacity at public hospitals in Zambia. Emerg Med J. 2019 Oct;36(10):620-624. doi: 10.1136/emermed-2018-207465. Epub 2019 Jul 10. PMID 31292206
- [Background] De Wulf A, Aluisio AR, Muhlfelder D, Bloem C. Emergency Care Capabilities in North East Haiti: A Cross-sectional Observational Study. Prehosp Disaster Med. 2015 Dec;30(6):553-9. doi: 10.1017/S1049023X15005221. Epub 2015 Oct 21. PMID 26487267
- [Background] Pigoga JL, Joiner AP, Chowa P, Luong J, Mhlanga M, Reynolds TA, Wallis LA. Evaluating capacity at three government referral hospital emergency units in the kingdom of Eswatini using the WHO Hospital Emergency Unit Assessment Tool. BMC Emerg Med. 2020 May 6;20(1):33. doi: 10.1186/s12873-020-00327-w. PMID 32375637
- [Background] Seo DH, Kim H, Kim KH, Park J, Shin DW, Park JM, Kim H, Jeon W, Kim JE. Status of Emergency Signal Functions in Myanmar Hospitals: A Cross-Sectional Survey. West J Emerg Med. 2019 Oct 24;20(6):903-909. doi: 10.5811/westjem.2019.7.43014. PMID 31738717
- [Background] Morse JM. The significance of standards. Qual Health Res. 2003 Nov;13(9):1187-8. doi: 10.1177/1049732303257231. No abstract available. PMID 14606408
- [Background] Guest G, Namey E, Chen M. A simple method to assess and report thematic saturation in qualitative research. PLoS One. 2020 May 5;15(5):e0232076. doi: 10.1371/journal.pone.0232076. eCollection 2020. PMID 32369511
- [Background] Guest G, Bunce A, Johnson L. How Many Interviews Are Enough?:An Experiment with Data Saturation and Variability. Field Methods. 2006;18(1):59-82. doi: 10.1177/1525822x05279903. 84. Guest G, MacQueen KM, Namey EE. Applied thematic analysis: Sage; 2012
- [Background] Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci. 2009 Aug 7;4:50. doi: 10.1186/1748-5908-4-50. PMID 19664226
- [Background] Kraemer HC, Mintz J, Noda A, Tinklenberg J, Yesavage JA. Caution regarding the use of pilot studies to guide power calculations for study proposals. Arch Gen Psychiatry. 2006 May;63(5):484-9. doi: 10.1001/archpsyc.63.5.484. PMID 16651505
- [Background] Chan CL, Leyrat C, Eldridge SM. Quality of reporting of pilot and feasibility cluster randomised trials: a systematic review. BMJ Open. 2017 Nov 8;7(11):e016970. doi: 10.1136/bmjopen-2017-016970. PMID 29122791
- [Background] Ardsby M, Shayo F, Sakita FM, Wilhelms D, Moshi B, Frankiewicz P, Silva LL, Staton CA, Mmbaga B, Joiner A. Emergency unit capacity in Northern Tanzania: a cross-sectional survey. BMJ Open. 2023 Feb 22;13(2):e068484. doi: 10.1136/bmjopen-2022-068484. PMID 36813501
- See also: A cohort of pediatric injury patients from a hospital-based trauma registry in Northern Tanzania — https://doi.org/10.1016/j.afjem.2022.04.008
- See also: WHO. Injuries and Violence: the facts 2014 [cited 2019 September 17] — https://apps.who.int/iris/bitstream/handle/10665/149798/9789241508018_eng.pdf?sequence=1
- See also: WHO. Basic emergency care: approach to the acutely ill and injured Geneva2018 [9/6/2022] — https://www.who.int/publications/i/item/basic-emergency-care-approach-to-the-acutely-ill-and-injured
- See also: Thaddeus S, Maine D. Too far to walk: Maternal mortality in context. Soc Sci Med. 1994;38(8):1091-110 — https://doi.org/10.1016/0277-9536(94)90226-7
- See also: Center FI. Fogarty-led project aims to advance emergency care research in low- and middle-income countries: National Institutes of Health, Department of Health and Human Services; 2019 [cited 2019 September 18] — https://www.fic.nih.gov/News/GlobalHealthMatters/july-august-2019/Pages/advancing-emergency-care-research-lmics.aspx
- See also: Eunice Kennedy Shriver National Institute of Child Health and Development. NICHD Strategic Plan 2020. Healthy pregnancies. Healthy children. Healthy and optimal lives.2020 October 4, 2022 — https://www.nichd.nih.gov/sites/default/files/2019-09/NICHD_Strategic_Plan.pdf

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-18): https://cdn.clinicaltrials.gov/large-docs/08/NCT06075108/Prot_SAP_000.pdf